CLINICAL TRIAL: NCT00100490
Title: Immune and Endocrine Function in Post-Traumatic Stress Disorder
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: CADE-RCD3
Record Dates: First submitted 2004-12-30; First posted 2004-12-31 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Post-Traumatic Stress Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This is a study investigating immune function and relationships to the hypothalamic-pituitary-adrenal (HPA) axis in Post-traumatic stress disorder (PTSD) compared to controls without PTSD. The study involves 99 adult veterans and civilian subjects over a 3 year period. The study involves measuring immune and neuroendocrine parameters from blood samples obtained before and after a dexamethasone suppression test. The aim of the study is to determine whether immune alterations exist in PTSD and whether the immune-HPA axis interactions in this disorder are different from non-PTSD subjects with the future aim of studying whether immune dysregulation in PTSD may be linked to the increased risk for medical and psychiatric comorbidity in this population.

DETAILED DESCRIPTION:
The subjects undergo a thorough medical (physical and blood/urine tests) and psychiatric evaluation to determine eligibility after signed informed consent is obtained. If eligible, the subject will complete questionnaires and undergo structured clinical interviews with a study psychiatrist. The subject will then undergo a 2-day testing period during which time, blood is drawn each morning at 8 am, with the subject taking 0.5 mg of dexamethasone (a synthetic steroid) at 11 pm prior to the second day of blood testing. About 80 ml of blood will be drawn on each morning. The blood collected will then be assayed for cortisol dexamethasone, lymphocyte glucocorticoid receptor levels; cytokine levels in plasma and lipopolysaccharide stimulated and unstimulated whole blood (IL-2, sIL-2R, IL-6, sIL-6R, and IL-10); lymphocyte subsets (T helper and suppressor, B, and Natural Killer cell numbers), and antigen stimulation responses to tetanus and candida. In addition, blood from the first day of testing will undergo ex vivo challenge with dexamethasone at varying concentrations to determine differential cytokine sensitivities to steroid exposure in subjects.

ELIGIBILITY:
* Subjects with DSM-IV criteria of PTSD and control subjects without any Axis I diagnosis, both groups of subjects are not on any psychotropic medications or medications that could interfere with the biological results, and do not have unstabilized medical conditions or neuroendocrine or immune disorders;
* Do not have comorbid psychosis, bipolar disorder, or substance use disorders;
* Have the capacity to give written informed consent;
* Do not have abnormalities on medical evaluation/physical examination;
* Are not a danger to self or others;
* Women subjects are not pregnant or lactacting, and use a safe form of contraception with a negative pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1999-10; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Yehuda, Ph.D.; Lloyd Mayer, M.D.; Esther Sternberg, M.D.; Bruce McEwen, Ph.D.
Locations (1):
- Bronx VAMC, The Bronx, New York, United States